CLINICAL TRIAL: NCT05928000
Title: Hellenic Multicenter Real-life Clinical Study for Bulevirtide Therapy in Chronic Hepatitis D: HERACLIS-BLV
Acronym: HERACLIS-BLV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Georgios Papatheodoridis, Professor Georgios Papatheodoridis, University of Athens
Other Study IDs: UAthens-HERACLIS-BLV
Record Dates: First submitted 2023-06-16; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Hepatitis D
Keywords: bulevirtide; NTCP inhibitor; Hepatitis D
MeSH Terms: conditions — Hepatitis D | interventions — bulevirtide; entecavir; Tenofovir; peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Serum samples for HDV RNA measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BLV-treated patients: All patients treated with daily Bulevirtide (BLV) subcutaneous injections of 2 mg, with or without concomitant use of a nucleos(t)ide analogue. Patients with concomitant use of pegylated interferon-alfa can be included.
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — BulevIrtide treatment in patients with chronic hepatitis D
  Other Names: Entecavir; Tenofovir; Pegasys

SUMMARY:
This study aims to assess the efficacy and safety of bulevirtide (BLV) in chronic hepatitis D patients treated in Greek liver centers.

DETAILED DESCRIPTION:
Background:

The prevalence of infection with hepatitis D virus (HDV) varies widely among different countries and even among different areas of the same country. Over the last decades, the prevalence of HDV infection was reported to be deceasing in most developed countries in parallel with the decreasing prevalence of chronic infection with hepatitis B virus (HBV). However, migration from countries with high HDV prevalence to countries with low HDV prevalence may have changed the HDV epidemiology in developed countries today. In Greece, the current prevalence of antibodies against HDV (anti-HDV) is approximately 5-6% among HBsAg-positive patients who visit the liver clinics of tertiary centers.

Regardless of HDV prevalence in any country, there is certainly underdiagnosis of HDV infection, since the majority of HBsΑg-positive cases are not screened for HDV. In particular in Greece, the anti-HDV screening rate of HBsAg-positive patients seen at tertiary liver centers does not exceed 50% having great variations among different centers.

It is well established that chronic HDV infection worsens the prognosis of HBsAg-positive patients increasing the risk of progression to cirrhosis and development of hepatocellular carcinoma (HCC). Therefore, there can be dramatic consequences if HDV patients are not diagnosed and thus are not properly managed. Until recently, pegylated interferon-alfa (pegIFNa) was the only agent that could be used for the treatment of patients with chronic hepatitis D. Given that pegIFNa has contraindications and suboptimal safety and tolerability profile, not all chronic hepatitis D patients could be treated or could remain on treatment. In addition, pegIFNa is not effective in all patients who can receive such treatment, whereas a large proportion of patients will experience relapses after the end of pegIFNa treatment.

In July 2020, the European Medicines Agency provided conditional approval for the use of bulevirtide (BLV) in patients with chronic hepatitis D. BLV inhibits the entry of HBV and consequently HDV in the hepatocytes by binding to and inactivating NTCP (Na+-taurocholate cotransporting polypeptide or sodium/bile acid cotransporter), which is a bile salt hepatocyte transporter also serving as HBV/HDV entry transporter by interacting with HBsAg. Due to the absence of effective treatment options for chronic hepatitis D, the approval of BLV was based only on data from phase ΙΙ trials including limited number of patients. Over the last two years, BLV has started to be used in limited countries including Greece and thus the systematic report of real life data on BLV in chronic hepatitis D is of great importance.

Aim:

The aim of this study is to assess the efficacy and safety of bulevirtide (BLV) in chronic hepatitis D patients treated in Greek liver centers.

Patients - Therapy:

This study will include all adult (>16 years old) patients with chronic hepatitis D followed at any of the participating centers who started BLV before the approval of the study protocol. Thus, the decision to use BLV will not be affected by the patient enrollment in the study, All patients will be treated with daily BLV subcutaneous injections of 2 mg, with or without concomitant use of a nucleos(t)ide analogue. Patients with concomitant use of pegylated interferon-alfa can be included.

Participating centers:

The following centers have been invited and agreed to participate in the HERACLIS-BLV study:

1. Department of Gastroenterology, Medical School of National & Kapodistrian University of Athens, General Hospital of Athens "Laiko";
2. 2nd Department of Internal Medicine, Medical School of National & Kapodistrian University of Athens, General Hospital of Athens "Hippokration";
3. Gastroenterology Department, General Hospital of Athens "Evangelismos";
4. 4th Department of Internal Medicine, General Hospital of Athens "Evangelismos";
5. University Department of Internal Medicine, General and Oncology Hospital of Kifisia "Agioi Anargyroi";
6. Gastroenterology Department, "Agios Savvas" General Anticancer-Oncology Hospital of Athens;
7. General Hospital Nikaia-Piraeus "Agios Panteleimon", General Hospital of Western Attica Agia Varvara;
8. Internal Medicine Department, 417 NIMTS (Army Equity Fund Hospital);
9. Gastroenterology Unit, General Hospital of Athens "Alexandra";
10. Liver Unit, Euroclinic SA, Athens;
11. Department of Medicine, and Research Laboratory of Internal Medicine, School of Medicine of University of Thessaly, University Hospital of Larissa;
12. 2nd Department of Internal Medicine, Aristotle University of Thessaloniki, General Hospital of Thessaloniki "Hippokratio";
13. 4th Department of Internal Medicine, Aristotle University of Thessaloniki, General Hospital of Thessaloniki "Hippokratio";
14. 1st Department of Internal Medicine, Democritus University of Thrace, Alexandroupolis;
15. Department of Gastroenterology, University Hospital of Patras;
16. Department of Gastroenterology, University Hospital of Ioannina;
17. Department of Gastroenterology & Hepatology, University Hospital of Heraklion Crete;
18. 1st Department of Internal Medicine, General Hospital of Rhodes, Greece.

Approvals:

Τhe protocol and the informed consent of this non-interventional study will be approved by the Ethical Committee of each participating hospital. All patients will sign an informed consent form.

Endpoints:

Primary

• Serum HDV RNA decline <2 log10 IU/ml and normal ALT at week 48

Secondary

* Serum HDV RNA decline <2 log10 IU/ml and normal ALT at week 96
* Undetectable serum HDV RNA at week 48
* Undetectable serum HDV RNA at week 96

Enrollment and study duration:

The enrollment period is expected to last 6 months; it is estimated that approximately 60-80 patients will be enrolled. The minimum follow-up will be 24 months after the onset of BLV, but non-final results will be available earlier. Final statistical analyses and manuscript preparation are expected to last 6 months. Thus, the total study duration is estimated to be 36 months.

Methods - Follow-up:

Patients' monitoring will be based on the principles of standard clinical practice according to the existing national recommendations for the treatment of patients with chronic hepatitis D. Thus, the patients' enrollment into this study will not affect the standard clinical practice for their management A predefined case report form (CRF) will be used for the collection of patients' data before the onset of BLV treatment. Then, standard clinic-laboratory data will be recorded at 6, 12, 18 and 24 months of BLV therapy. The patients' data at different visits will be recorded retrospectively or prospectively depending on the duration of BLV at their inclusion in this study.

Statistical analysis:

All data will be recorded in a specifically designed CRF and will be entered into a specifically designed Excel form and then SPSS database for analyses.

ELIGIBILITY:
Inclusion Criteria:

* All adult (>16 years old) patients with chronic hepatitis D followed at any of the participating centers
* Start of BLV treatment before the approval of the study protocol.
* Any patient with or without concomitant use of a nucleos(t)ide analogue. Patients with concomitant use of pegylated interferon-alfa can be included.

Exclusion Criteria:

* Any patient with chronic hepatitis D who started BLV after the start of the study protocol

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include all adult (>16 years old) patients with chronic hepatitis D followed at any of the participating centers who started BLV before the approval of the study protocol. Thus, the decision to use BLV will not be affected by the patient enrollment in the study,
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Response at week 48 | Week 48
  Proportion of patients with serum HDV RNA decline >=2 log10 IU/ml and normal ALT

SECONDARY OUTCOMES:
Response at week 96 | Week 96
  Proportion of patients with serum HDV RNA decline >=2 log10 IU/ml and normal ALT
Complete response at week 48 | Week 48
  Proportion of patients with undetectable serum HDV RNA
Complete response at week 96 | Week 96
  Proportion of patients with undetectable serum HDV RNA

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Medical School of National & Kapodistrian University of Athens, General Hospital of Athens "Laiko";, Athens, Greece

REFERENCES:
- [Result] Papatheodoridi M, Papatheodoridis GV. Is hepatitis delta underestimated? Liver Int. 2021 Jun;41 Suppl 1:38-44. doi: 10.1111/liv.14833. PMID 34155795
- [Result] Wedemeyer H. The burden of hepatitis D - defogging the epidemiological horizon. J Hepatol. 2020 Sep;73(3):493-495. doi: 10.1016/j.jhep.2020.06.037. Epub 2020 Jul 16. No abstract available. PMID 32684365
- [Result] Papatheodoridis G, Mimidis K, Manolakopoulos S, Triantos C, Vlachogiannakos I, Veretanos C, Deutsch M, Karatapanis S, Goulis I, Elefsiniotis I, Cholongitas E, Sevastianos V, Christodoulou D, Samonakis D, Manesis E, Kapatais A, Papadopoulos N, Ioannidou P, Germanidis G, Giannoulis G, Lakiotaki D, Kogias D, Kranidioti Eta, Zisimopoulos K, Mela M, Kontos G, Fytili P, Manolaka C, Agorastou P, Pantzios SI, Papatheodoridi M, Karagiannakis D, Geladari E, Psychos N, Zachou K, Chalkidou A, Spanoudaki A, Thomopoulos K, Dalekos G. HERACLIS-HDV cohort for the factors of underdiagnosis and prevalence of hepatitis D virus infection in HBsAg-positive patients. Liver Int. 2023 Sep;43(9):1879-1889. doi: 10.1111/liv.15638. Epub 2023 Jun 8. PMID 37288712
- [Result] Papatheodoridi M, Papatheodoridis GV. Current status of hepatitis delta. Curr Opin Pharmacol. 2021 Jun;58:62-67. doi: 10.1016/j.coph.2021.03.008. Epub 2021 Apr 22. PMID 33895531
- [Result] Bogomolov P, Alexandrov A, Voronkova N, Macievich M, Kokina K, Petrachenkova M, Lehr T, Lempp FA, Wedemeyer H, Haag M, Schwab M, Haefeli WE, Blank A, Urban S. Treatment of chronic hepatitis D with the entry inhibitor myrcludex B: First results of a phase Ib/IIa study. J Hepatol. 2016 Sep;65(3):490-8. doi: 10.1016/j.jhep.2016.04.016. Epub 2016 Apr 27. PMID 27132170
- [Result] Wedemeyer H, Aleman S, Brunetto MR, Blank A, Andreone P, Bogomolov P, Chulanov V, Mamonova N, Geyvandova N, Morozov V, Sagalova O, Stepanova T, Berger A, Manuilov D, Suri V, An Q, Da B, Flaherty J, Osinusi A, Liu Y, Merle U, Schulze Zur Wiesch J, Zeuzem S, Ciesek S, Cornberg M, Lampertico P; MYR 301 Study Group. A Phase 3, Randomized Trial of Bulevirtide in Chronic Hepatitis D. N Engl J Med. 2023 Jul 6;389(1):22-32. doi: 10.1056/NEJMoa2213429. Epub 2023 Jun 22. PMID 37345876